CLINICAL TRIAL: NCT03601975
Title: Phase III Randomized Trial of Anlotinib Plus Gemcitabine/Cisplatin Vesus Placebo Plus Gemcitabine/Cisplatin in Previous Untreated Patients With Recurrent/Metastatic Nasopharyngeal Carcinoma
Brief Title: Gemcitabine and Cisplatin With/Without Anlotinib in Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALTN-17-III
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anlotinib plus Gemcitabine/Cisplatin (Experimental): patients receive anlotinib at 12mg QD (d1-d14)and gemcitabine (1000 mg/m² d1,8) or cisplatin (80mg/m² d1) every 3 weeks for every cycle
  Interventions: Drug: Gemcitabine/Cisplatin
- placebo plus Gemcitabine/Cisplatin (Placebo Comparator): patients receive pacebo at 0mg QD (d1-d14)and gemcitabine (1000 mg/m² d1,8) or cisplatin (80mg/m² d1) every 3 weeks for every cycle
  Interventions: Drug: Gemcitabine/Cisplatin

INTERVENTIONS:
Drug: Gemcitabine/Cisplatin — gemcitabine (1000 mg/m² d1,8) or cisplatin (80mg/m² d1) every 3 weeks for every cycle

SUMMARY:
This is a Phase III randomized controlled multi-center trial comparing anlotinib plus Gemcitabine/Cisplatin with placebo plus Gemcitabine/Cisplatin in previous untreated patients with recurrent/metastatic Nasopharyngeal Carcinoma, in order to verify the efficacy and security of anlotinib in mNPC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Informed of the investigational nature of this study and give written informed consent
2. Histologically or cytologically confirmed nasopharyngeal carcinoma, tumor staged as IVB (according to the 8th AJCC edition) or recurrent tumor nott suitable for local treatment.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 to1, life expectancy of at least 12 weeks.
4. Antitumor therapy naive for recurrent or metastatic nasopharyngeal carcinoma
5. Completed radiotherapy for local tumor 4 weeks before the enrollment
6. Measurable disease other than brain metastasis based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
7. Adequate organ system function, defined as follows:

   1. ANC ≥1.5×109/L, PLT ≥100×109/L, Hb）≥90g /L;
   2. TBIL ≤ 1.5×ULN；Aminopherases (ALT and AST) ≤ 2.5 × ULN (without liver metastasis) or ≤ 5.0 × ULN (with liver metastasis), Creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 ml/min;
   3. Urine protein < ++，or urine protein ≥ ++ concomitant with content of -hour urinary protein <1.0 g;
   4. INR≤1.5×ULN, APTT≤1.5×ULN;
   5. LVEF ≥50%;
8. Women who are not of child-bearing potential, and women of child-bearing potential who have a negative serum or urine pregnancy test prior to initial trial treatment, and who agree to use adequate contraceptive measures during the study; Men with partners of childbearing potential willing to use adequate contraceptive measures during the study

Exclusion Criteria:

1. Patients with a previous malignancy within the past 5 years (other than curatively treated in situ carcinoma of the cervix, non-melanoma skin cancer and superficial bladder carcinoma).
2. Allergic to anotinib or the chemotherapeutic agents involved in this trial;
3. Supposed to receive locally treatment (except for those with symptomatic bone metastases receive appropriate local doses radiotherapy which does not affect the hemogram)
4. Patients that have received definitive radiotherapy, adjuvant chemotherapy or cocurrent chemoradiotherapy for stage I-IVA and developed recurrent disease within 6 months;
5. Patients that have previously received target therapies;
6. Patients that have previously received immunotherapy (i.e.,interferon, or IL-2 ) 28 days before randomization or within 5 half-life of the drug.
7. Patients that have previously received immunosupressive drugs (i.e., Corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide or TNF-α)
8. Symptomatic CNS metastasis (i.e. encephaledema, hormone intervention, or brain metastasis progression)
9. Patients currently have bleeding tendency, including but not limited to gastrointestinal bleeding, nasal bleeding, hemoptysis, and persistent bleeding or coagulopathy;
10. Hemoptysis (defined as coughing out or spitting out ≥ 1 teaspoon of blood or small blood clots or hemoptysis without sputum) within 28 days before randomization, not including bloody sputum.
11. Radiograph (within 28 days before randomization) showed that the tumor surrounded important blood vessels, and the investigators determined that entering the study would cause bleeding risk;
12. Subjects have any of the following severe acute complications:

    1. Unstable angina and/or congestive heart failure or vascular disease (eg, aortic aneurysm requires surgically repaired or peripheral venous thromboembolism) requiring hospitalization within 12 months, or other cardiac impairments (eg,uncontrolled arrhythmias) determined by the investigator, which may affect the evaluation of drug safety; Myocardial infarction or ischemia with ST elevation ≥ 2 mm indicated by ECG;
    2. Arterial thromboembolism, venous thromboembolism in grade 3 or higher (according to NCI-CTCAE), transient ischemic attack (TIA), cerebral vascular accident (CVA), transmural myocardial infarction ( MI), hypertensive crisis or hypertensive encephalopathy within 24weeks;
    3. Chronic Obstructive Pulmonary Disease (COPD) or other respiratory diseases requiring hospitalization within 28 days before randomization;
    4. Abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, or acute gastrointestinal bleeding within 24 weeks before randomization;
    5. Esophageal and gastric varices, unhealed ulcers, unhealed wounds or fracture within 24 weeks before randomization;
    6. Pulmonary infections and/or acute bacterial or fungal infections requiring intravenous antibiotic therapy
    7. Clinical jaundice and/or coagulation disorders caused by liver dysfunction;
    8. Minor surgical procedures (including catheterization, excluding peripheral venipuncture central vena catheterization) within 2 days of randomization;
13. The virological test indicates that either of the following 28 days before randomization

    1. HBsAg positive and HBV DNA ≥ 1 × 103 copies/L;
    2. Anti-HCV positive
    3. HIV positive
14. Participation of an anti-tumor clinic trial within 28 days before randomization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2018-08-27 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 12months
  Progeression free survival is calculated from randomization to disease progeression or death

CONTACTS AND LOCATIONS:
Locations (1):
- 651 Dongfeng Road East, Yuexiu District, Guanzhou, P.R. China, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No